CLINICAL TRIAL: NCT01180556
Title: The Effect of Probiotics in Childhood Abdominal Pain
Brief Title: Effect of Probiotics in Childhood Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sor493009ctil; 4930 (Other: SMC)
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Pain
Keywords: childhood; abdominal pain; probiotics
MeSH Terms: conditions — Abdominal Pain | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics supplementation (Experimental): Supplementation by probiotics for 4 weeks
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Supplementation of placebo for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Daily oral supplementation for four weeks
  Other Names: probiotic agent, L. reuteri
  Arms: Probiotics supplementation
Dietary Supplement: Placebo — Placebo administration
  Other Names: placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of probiotics in childhood recurrent abdominal pain. Patients will be randomly assigned to receive L. reuteri or placebo for 4 weeks with a follow up phase of additional 4 weeks.

DETAILED DESCRIPTION:
Prospective randomized double-blind placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children

Exclusion Criteria:

* Any chronic or organic illness

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of abdominal pain | Eight weeks
  Number of pain episodes and pain intensity based on a visual scale

SECONDARY OUTCOMES:
School absenteeism | Eight weeks
  Number of patients with school absenteeism
Other gastrointestinal symptoms | Eight weeks
  Any gastrointestinal symptom such as nausea, vomiting, diarrhea, bloating
Adverse effects related to treatment | Eight weeks
  Any adverse effects related to the probiotic supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Weizman, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weizman Z, Abu-Abed J, Binsztok M. Lactobacillus reuteri DSM 17938 for the Management of Functional Abdominal Pain in Childhood: A Randomized, Double-Blind, Placebo-Controlled Trial. J Pediatr. 2016 Jul;174:160-164.e1. doi: 10.1016/j.jpeds.2016.04.003. Epub 2016 May 4. PMID 27156182